CLINICAL TRIAL: NCT03806478
Title: Safety, Tolerability and Efficacy Assessment of Intranasal Nanoparticles of APH-1105, A Novel Alpha Secretase Modulator For Mild to Moderate Cognitive Impairment Due to Alzheimer's Disease(AD)
Brief Title: Study of APH-1105 in Patients With Mild to Moderate Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aphios (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APH-1105
Record Dates: First submitted 2019-01-04; First posted 2019-01-16 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Dementia; Alzheimer Disease 1; Alzheimer Disease 2; Alzheimer Disease 3
Keywords: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Dementia; Alzheimer disease type 1; Alzheimer disease type 2; Alzheimer disease, familial, type 3; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Exploratory Phase 2 Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 0.5 µg (Experimental): Intranasal (IN) nanoparticles - 0.5 micrograms. The study is planned to include 1 dose of APH 1105 / 0.5 µg, administered twice a week for 12 weeks, for a total of 24 doses.
  Interventions: Drug: APH-1105
- 1.0 µg (Experimental): Intranasal (IN) nanoparticles - 1.0 micrograms. The study is planned to include 1 dose of APH 1105 / 1.0 µg, administered twice a week for 12 weeks, for a total of 24 doses.
  Interventions: Drug: APH-1105
- 2.0 µg (Experimental): Intranasal (IN) nanoparticles - 2.0 micrograms. The study is planned to include 1 dose of APH 1105 / 2.0 µg, administered twice a week for 12 weeks, for a total of 24 doses.
  Interventions: Drug: APH-1105
- Placebo (Placebo Comparator): Intranasal (IN) Placebo nanoparticles. The study is planned to include 1 dose of placebo drug administered twice a week for 12 weeks, for a total of 24 doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: APH-1105 — The investigational drug product, APH-1105 is a sterile, pyrogen-free lyophilized powder intended for intranasal administration.
  Arms: 0.5 µg; 1.0 µg; 2.0 µg
Other: Placebo — The placebo is a sterile, pyrogen free lyophilized powder identical in appearance to the experimental drug
  Arms: Placebo

SUMMARY:
This is a Phase 2 study assessing the safety, tolerability and efficacy of intranasal delivery of APH-1105 for the treatment of mild to moderate Alzheimer's in adult.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, triple blind placebo-control with parallel groups. Patients diagnosed with mild to moderate AD will be enrolled and randomly assigned in a blinded fashion to receive study drug APH-1105. Groups will receive either 0.5 µg (15 active, 5 placebo), 1.0 µg (15 active, 5 placebo), or 2.0 µg (15 active, 5 placebo). A full assessment will be made of all relevant tolerability and safety data.

Patients will be administered the study drug outside of the clinic setting by a study partner twice a week. The initial dose of APH-1105 will take place in a clinic setting for the purpose of collecting initial Pharmacokinetic data.

The total duration for patient participation will be approximately 18 weeks which includes 1 week for screening, 12 weeks of treatment and followup 4 weeks post final dose. Study visits will occur during screening, baseline, weeks 1, 2, 4, 8, 12 and 16 for a total of 7 visits. Week 16 represents the followup visit after the final dose of study medication.

Cognitive assessments will be performed at screening, and will repeat at weeks 4, 12 and 16. Behavioral Functioning and Quality of Life measures will be done at weeks 2,4,8,12 and 16.

Blood samples will collected though out the study for Pharmacokinetic analyses.

ELIGIBILITY:
Inclusion Criteria

* Males and Females ages > 50 years of age at screening visit
* Probable Alzheimer's Disease according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association(NINCDS-ADRDA) and Diagnostic Statistical Manual (DSM) IV-V criteria
* Clinical Dementia Rating Scale (CDR) global score > 1.0 at the time of screening
* Mini-Mental Status Examination score of 22-30 at screening visit CT or MRI of brain, within 12 months prior to randomization, compatible with a diagnosis of Probable Alzheimer's Disease
* Physical examination, laboratory data and electrocardiogram results from screening visit must be normal or abnormal findings must be judged not to be clinically significant
* Ability to walk, at least with an assistive device
* Vision and hearing sufficient to comply with testing
* Informed consent from patient, or legal guardian (if applicable) and a caregiver
* Living outside an institutional facility
* Must have at least 1 informant/study partner

Exclusion Criteria

* Clinically significant and active pulmonary, gastrointestinal, renal, hepatic, endocrine or cardiovascular system diseases
* Other neurological disorders, including but not limited to stroke, Parkinson's Disease, seizure disorder, or head injury with loss of consciousness within the past 5 years
* DSM-IV Axis I disorder other than Alzheimer's Disease, including amnesic disorders, schizophrenia or schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic, or post-traumatic stress disorder
* CT scan or MRI evidence of hydrocephalus, stroke, a space-occupying lesion, cerebral infection, or any other clinically significant central nervous system disease
* Dementia complicated by another organic disease
* Dementia complicated by the presence of predominant delusions
* Patients with a hematological malignancy or solid tumor who are undergoing treatment, who have completed treatment within the past 6 months, or who still have evidence of active disease
* Current drug or alcohol dependency including nicotine addiction (smokers)
* Subjects receiving immune-suppressants tricyclic antidepressants anticoagulants or chemotherapeutic agents
* Hypertension that is poorly controlled or managed
* Any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns
* Clinically significant, unstable psychiatric illness
* Have had a stroke or Transient Ischemic Attack (TIA) or unexplained loss of consciousness in the past 1 year
* Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
* History of unstable angina, myocardial infarction, chronic heart failure or clinically significant conduction abnormalities within 1 year prior to Screening Visit 1
* Indication of impaired renal or liver function
* Clinically significant systemic illness or serious infection within 30 days prior to or during the screening period
* Use of allowed medications for chronic conditions at doses that have not been stable for at least 4 weeks prior to Screening Visit 1, or use of AD medications at doses that have not been stable for at least 8 weeks prior to Screening Visit 1
* Use of any medications that, in the opinion of the Investigator, may contribute to cognitive impairment, put the participants at higher risk for adverse events (AEs), or impair the participant's ability to perform cognitive testing or complete study procedures.
* Contraindications to study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of Treatment-emergent Adverse Events | Baseline through 30 days post final treatment dose up to day 60
  Number of patients experiencing Adverse (AE) and Serious Adverse (SAE) events during treatment and followup.
Efficacy: Cognition Change | Baseline - day 60
  Change in Alzheimer's Disease Assessment Scale-Cog (ADAS-COG) total score from baseline to post final treatment dose.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale test(ADAS-Cog) measures language and memory and is comprised of 2 parts targeting cognitive and non-cognitive functioning. It consists of 11 items which include (but not all) word recall, naming of objects, word recognition, comprehension and word finding. The ADAS-COG is scored 0-70. The higher the score the greater the impairment.
Efficacy: Change in Cognitive Functioning | Baseline - day 60
  Change in the Hopkins Verbal Learning Test-Revised from baseline to day 60 post final treatment dose The Hopkins Verbal Learning Test, a three-trial list of 12 words is a learning and free recall task. The Hopkins Verbal Learning Test measures episodic memory. The test is made up of three trials which requires the patient to free-recall words from the 12 word list involving yes/no responses. The score range is from 0-12. Lower scores (numbers) indicate more impairment.

SECONDARY OUTCOMES:
Tolerability: [Pharmacokinetics] Cmax | Blood draws at baseline and 15 minutes, 30minutes, 60minutes, 2 hours, 6hours, 12hours, 24hours, 48hours and 72hours post first administered dose
  Characterize pharmacokinetic effects of APH-1105 exposure in patients with Alzheimer's Disease to determine peak plasma concentration (Cmax).
Tolerability: [Pharmacokinetics] Tmax | Blood draws at baseline and 15 minutes, 30minutes, 60minutes, 2 hours, 6hours, 12hours, 24hours, 48hours and 72hours post first administered dose
  Characterize pharmacokinetic effects of APH-1105 exposure in patients with Alzheimer's Disease to determine peak serum concentration(Tmax).
Tolerability: [Pharmacokinetics] serum elimination half life | Blood draws at baseline and 15 minutes, 30minutes, 60minutes, 2 hours, 6hours, 12hours, 24hours, 48hours and 72hours post first administered dose
  Characterize pharmacokinetic effects of APH-1105 exposure in patients with Alzheimer's Disease to determine serum elimination half life(1/2).
Tolerability: [Pharmacodynamics] protein kinase C activity | Blood draws at baseline, 15 minutes, 30minutes, 60minutes, 2hours, 6hours, 12hours, 24hours, 48hours, and 72hours post first administered dose.
  Assess the Protein Kinase C Activity in patients treated with multiple doses of APH-1105
Change in Behavioral Functioning | Baseline, week 4, 8 12 and week 16 post final dose.
  Change in the Behavioral Pathology in Alzheimer's Disease Rating Scale -Frequency-Weighted (BEHAVE-AD-FW). The Behavioral Pathology in Alzheimer's Disease Frequency Weighted Severity Scale (BEHAVE-AD-FW) assesses the possible neurological basis of behavioral and psychological symptoms of dementia, the relationships between behavioral functioning and cognitive functioning. The scale consists of seven (7) behavioral categories (paranoid and delusional ideation, hallucinations, activity disturbances, aggressiveness, diurnal rhythm disturbances, affective disturbances, anxieties, and phobias) and consists of twenty-five (25) symptoms grouped into these categories. Items are score on a 4 point severity - higher the score, higher the impairment.
Change in Behavioral Disturbance | Baseline, week 4, 8 12 and week 16 post final dose.
  Change in the Neuropsychiatric Inventory (NPI) The Neuropsychiatric Inventory (12 item) is a caregiver/informant-based interview that assesses 12 neuro-psychiatric symptoms of the participant over the previous month. Responses are rated both in terms of frequency (1=rarely, less than once per week; 2=sometimes, about once per week; 3=often, several times per week; and 4=very often, once or more per day) and severity (1=mild; 2=moderate; 3=severe) with composite scores ranging from 0-144. The higher the score the greater symptom severity.
Change in Dementia Symptom Severity | Baseline, week 4, 8 12 and week 16 post final dose.
  Change in the Clinical Dementia Rating Scale(CDR_SB) The Clinical Dementia Rating or CDR measure the stage severity of dementia. It is a five-point scale in which "0" connotes no cognitive impairment, and then the remaining four points are for various stages of dementia, mild to severe.
Evaluate the Quality of Life Status | Baseline, week 4, 8, 12 and week 16 post final dose
  Change in the Clinical Global Impression of Improvement (CGI-I) and the Caregiver Clinical Global Impression of Improvement (CGI-I) is a 3-item observer-rated scale that measures illness severity, global improvement or change, and therapeutic response. It is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse). Each component of the CGI is rated separately; the instrument does not yield a global score.
Risk of Suicide | Baseline, week 4, 8, 12 and week 16 post final dose
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. It is comprised of ten categories, with binary responses (yes/no) to indicate a presence or absence of the behavior. The ten categories included in the C-SSRS are as follows: Category 1 - Wish to be Dead; Category 2 - Non-specific Active Suicidal Thoughts; Category 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Category 5 - Active Suicidal Ideation with Specific Plan and Intent; Category 6 - Preparatory Acts or Behavior; Category 7 - Aborted Attempt; Category 8 - Interrupted Attempt; Category 9 - Actual Attempt (non-fatal); Category 10 - Completed Suicide. A yes/no binary response is also utilized in assessing self-injurious behavior without suicidal intent. The outcome of the C-SSRS is a numerical score obtained from the these categories.

IPD SHARING:
Plan to Share IPD: No